CLINICAL TRIAL: NCT00217854
Title: Mechanisms of Airway Inflammation: Natural Exacerbation of Asthma Induced by Glucocorticoid Withdrawal
Brief Title: Inflammatory Processes in the Airway of Asthmatics With Persistent Bronchial Hyperreactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mario Castro, Professor of Medicine and Pediatrics, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 291; P50HL056419 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: asthma, corticosteroids
MeSH Terms: conditions — Asthma

ARMS (1):
- Open label inhaled fluticasone (Other): Patients are treated with open label high dose fluticasone for 30 days then discontinued. Comparisons are pre- and post- treatment single arm.
  Interventions: Procedure: Bronchoscopic

INTERVENTIONS:
Procedure: Bronchoscopic — Bronchoscopic procedure

SUMMARY:
The purpose of this study is to examine inflammatory processes in the airway of moderate to severe persistent asthmatics who have persistent bronchial hyperreactivity despite chronic administration of inhaled glucocorticoids.

DETAILED DESCRIPTION:
BACKGROUND:

The Inhaled Glucocorticoid Withdrawal Protocol will investigate abnormalities in the asthmatic airway that occur in the setting of a "natural" endogenous exacerbation. It is known that chronic treatment with inhaled glucocorticoids causes a nearly complete disappearance of inflammatory cells from the airway and improvement in bronchial hyperreactivity, yet such patients have persistent bronchial hyperreactivity. Withdrawal of inhaled glucocorticoids causes a worsening of bronchial hyperreactivity. These observations suggest that a chronic derangement in the asthmatic airway might exist, which is unmasked by withdrawal of inhaled glucocorticoids and which reinitiates the inflammatory process. These "persistent" abnormalities in the asthmatic airway may be seen during quiescent stages of chronic asthma even when airway inflammatory changes are not evident. The abnormalities may be seen during the period of treatment with inhaled glucocorticoids or they may appear as one of the first signs after the withdrawal of inhaled glucocorticoids, thereby initiating the recurrence of asthma and promoting inflammation.

DESIGN NARRATIVE:

The purpose of this study is to examine inflammatory processes in the airway of moderate to severe persistent asthmatics who have persistent bronchial hyperreactivity despite chronic administration of inhaled glucocorticoids. Each participant will undergo bronchoscopic procedures and have assessment of bronchial hyperreactivity at the following two time points: 1) during treatment with inhaled fluticasone; and 2) after acute withdrawal of inhaled fluticasone.

The primary outcome of this study is the change in CD3 positive T cells in the airway submucosa.

The key secondary outcomes are as follows: 1) other inflammatory cell markers in the airway (e.g., CD4, CD8, CD68, CD45, EG2/MBP, tryptase, and neutrophil elastase); 2) RANTES (regulated on activation, normal T expressed and secreted) expression in airway; 3) FEV1 peak expiratory flows; 4) methacholine PC20; and 5) asthma symptom score.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of asthma as defined by the American Thoracic Society (ATS) definition. This includes the following:

  1. history of episodic shortness of breath (with or without associated wheezing) in association with reversible obstructive airways disease with at least a 20% decrement in FEV1 and FVC (from predicted values) that is documented at some time point by pulmonary function tests
  2. an improvement in expiratory flow rates of at least 15% of predicted values after inhalation of a beta-2 selective bronchodilator medication or other previous treatment (e.g. corticosteroids)
* The diagnosis may also be confirmed by an abnormal bronchospastic response to methacholine or exercise as described by Cherniak
* FEV1 greater than or equal to 70% of predicted value at time of study entry
* Regular use of inhaled corticosteroids at time of study entry (at least 400 mcg of Beclomethasone or equivalent)

Exclusion Criteria:

* Used inhaled cromolyn (Intal) or nedocromil (Tilade) in the month prior to study entry
* History of severe asthma requiring intubation
* Any cardiopulmonary or neurologic abnormality with which the risk of performing the procedure would outweigh the potential benefits (other than asthma)
* Upper respiratory tract infection or clinical evidence of a sinus infection during the month preceding the test
* History of cigarette smoking within the 5 years prior to study entry or greater than 10 pack-years total
* Pregnant or refuses to undergo urine pregnancy testing if female of child-bearing age (women of childbearing potential will not be challenged [methacholine challenge] unless they have had a menstrual period in the last 10 days or a negative pregnancy test within 2 weeks or are practicing adequate contraception)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2001-09; Primary Completion 2009-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
change in CD3 positive T cells in the airway submucosa | Measured at Week 4

SECONDARY OUTCOMES:
inflammatory cell markers in the airway (CD4, CD8, CD68, CD45, EG2/MBP, tryptase, and neutrophil elastase) | Measured at Week 4
RANTES expression in airway | Measured at Week 4
FEV1, peak expiratory flows | Measured at Week 4
methacholine PC20 | Measured at Week 4
asthma symptom score | Measured at Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Mario Castro, Study Chair — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Castro M, Bloch SR, Jenkerson MV, DeMartino S, Hamilos DL, Cochran RB, Zhang XE, Wang H, Bradley JP, Schechtman KB, Holtzman MJ. Asthma exacerbations after glucocorticoid withdrawal reflects T cell recruitment to the airway. Am J Respir Crit Care Med. 2004 Apr 1;169(7):842-9. doi: 10.1164/rccm.200208-960OC. Epub 2004 Jan 15. PMID 14726420
- See also: Click here for the Pulmonary and Critical Care Medicine Website — http://pulmonary.wustl.edu/